CLINICAL TRIAL: NCT04692298
Title: Pulse Consumption Improves Gut Health, Metabolic Outcomes, and Bone Biomarkers of Postmenopausal Women
Brief Title: Effects of Pulse Consumption on Bone Health of Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Edralin Lucas, Jim an Lynn Williams Professor, Oklahoma State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-20-430
Record Dates: First submitted 2020-12-16; First posted 2020-12-31 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Menopause
Keywords: bone health; pulses; microbiome
MeSH Terms: interventions — Pulse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulse (Other): Participants will consume kidney beans, lentil, pinto beans, black-eyed pea, chickpea
  Interventions: Other: pulses

INTERVENTIONS:
Other: pulses — kidney beans, pinto beans, lentil, black-eyed pea and chickpea

SUMMARY:
This study will investigate the effects of the addition of 100 grams/day of cooked pulses (i.e. lentil, pinto beans, peas, chickpeas, kidney beans) to the diet of postmenopausal women for 12 weeks on gut health, metabolic outcomes and bone biomarkers.

DETAILED DESCRIPTION:
With approximately 1.3 million women reaching menopause each year in the US and about one-third of a woman's life is spent in this state, it is imperative to identify effective, safe, and economical approaches that can minimize disease risk that is associated with this phase of life. Pulses are excellent source of fiber, protein, essential amino acids, vitamins, minerals and phytochemicals, that can act as prebiotics and prevent gut dysbiosis and promote a healthy gut. A few studies in overweight or obese adults have shown the health benefits of pulses, including gut modulating potential. However, studies examining the use of pulse crops are limited, especially in alleviating health risks associated with menopause. The objective of this study is to evaluate the prebiotic potential of pulse-based diet and consequent effects on metabolic and bone biomarkers in postmenopausal women. We hypothesize that daily intake of pulses, due to its nutrient content and many other bioactive compounds including fiber content, will beneficially affect gut health and subsequently improve metabolic outcomes and bone markers in postmenopausal women. To accomplish our objectives, 40 postmenopausal women (50- 65 y old and ≥ 1 y menopause) will be recruited and will be asked to consume 100 g/d of pulse (alternate between lentils, pinto beans, peas, chickpeas, and kidney beans) for 3 months. Pulse intake, anthropometric measures, markers of gut and bone health, and metabolic outcomes will be assessed at baseline and at the end of pulse consumption.

Once the study was underway and we got more funding, women were given the option to continue pulse supplementation for another six months to examine changes on bone density.

ELIGIBILITY:
Inclusion Criteria:

* 1 year without menstrual cycle

Exclusion Criteria:

* any medication use (for the past 6 m) that affects glucose, lipids, bone and inflammation markers, dietary supplements, and non-steroidal anti-inflammatory medications
* allergy to pulse crops
* tobacco use
* excessive alcohol intake
* antibiotic use
* major surgery within 6 m of study enrollment

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 41 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
changes in blood biomarkers and/or bone mineral density (BMD) | change from baseline, after 90 days and 9 months (for BMD)
  analyzed by enzyme linked immunoassay or dual energy xray absorptiometry for BMD
blood C-terminal telopeptide of type 1 collagen (CTX) | change from baseline after 90 days
  analyzed by enzyme-linked immunoassay
blood procollagen type 1 N-propeptide (P1NP) | change from baseline after 90 days
  analyzed by enzyme-linked immunoassay
fecal bacteria | change from baseline after 90 days
  analyzed by 16sRNA sequencing
fecal short chain fatty acid | change from baseline after 90 days
  analyzed by gas chromatography
fecal immunoglobulin A | change from baseline after 90 days
  analyzed by enzyme-linked immunoassay
plasma concentrations of fatty acid binding protein | change from baseline after 90 days
  analyzed by enzyme-linked immunoassay

SECONDARY OUTCOMES:
fasting blood glucose | change from baseline after 90 days
  analyzed using clinical chemistry analyzer
blood glycosylated hemoglobin | change from baseline after 90 days
  analyzed using clinical chemistry analyzer
blood insulin | change from baseline after 90 days
  analyzed using enzyme linked immunoassay
blood C-peptide | change from baseline after 90 days
  analyzed using enzyme linked immunoassay
blood total cholesterol | change from baseline after 90 days
  analyzed using clinical chemistry analyzer
blood HDL cholesterol | change from baseline after 90 days
  analyzed using clinical chemistry analyzer
blood LDL cholesterol | change from baseline after 90 days
  analyzed using clinical chemistry analyzer
blood triglycerides | change from baseline after 90 days
  analyzed using clinical chemistry analyzer

CONTACTS AND LOCATIONS:
Overall Officials: EDRALIN A LUCAS, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Nutritional Sciences Department, Oklahoma State University, Stillwater, Oklahoma, United States